CLINICAL TRIAL: NCT07385248
Title: An Open-label, Randomized, 2-treatment, 2-sequence, 2-period, Crossover Study to Evaluate the Pharmacokinetics and Safety Between the Administration of AD-229 and the Administration of AD-2291 for Healthy Adults in Fasting State
Brief Title: A Clinical Trial to Assess the Pharmacokinetics and Safety of AD-229 Compared to AD-2291 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-229BE
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1 : Reference Drug(AD-2291), Period 2 : Test Drug(AD-229)
  Interventions: Drug: AD-229; Drug: AD-2291
- Sequence B (Experimental): Period 1 : Test Drug(AD-229), Period 2 : Reference Drug(AD-2291)
  Interventions: Drug: AD-229; Drug: AD-2291

INTERVENTIONS:
Drug: AD-229 — AD-229 Oral Tablet
Drug: AD-2291 — AD-2291 Oral Tablet

SUMMARY:
The study compare and evaluate the safety and pharmacokinetic characteristics between the administration of AD-229 and the administration of AD-2291 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 kg/m2 and 29.9 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit

Exclusion Criteria:

* Participation in another clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration of drug in plasma (Cmax) | pre-dose (0hour) to 72hours
  Cmax of AD-229
Area under the plasma concentration-time curve during dosing interval (AUCt) | pre-dose (0hour) to 72hours
  AUCt of AD-229

IPD SHARING:
Plan to Share IPD: No